CLINICAL TRIAL: NCT06694597
Title: Efficacy and Safety of Astragalus Membranaceus on the Improvement of Cognitive and Non-cognitive Symptoms in Mild-to-Moderate Alzheimer's Disease
Brief Title: Efficacy, Safety of Astragalus Membranaceus in Mild-to-Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Huangqi_AD
Record Dates: First submitted 2024-09-04; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Huang Qi

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Astragalus membranaceus (Experimental)
  Interventions: Drug: Astragalus Membranaceus Root
- Routine treatment (No Intervention)

INTERVENTIONS:
Drug: Astragalus Membranaceus Root — Astragalus tablets 15g, warm water to drink, once a day, take for 1 year, during which routine treatment should also be carried out.
  Arms: Astragalus membranaceus

SUMMARY:
Alzheimer's disease (AD), the most common cause of dementia, is characterized by cognitive impairment, mental and behavioural abnormalities, and social dysfunction. Current treatments can only delay the progression of AD, not cure it completely. In vitro studies have shown that Astragalus has toxic effects such as anti-hypoxia injury of nerve cells, anti-free radical damage, anti-excitatory amino acids, etc. It can be used to expand cerebral vessels, increase cerebral blood flow, improve cerebral microcirculation, protect brain cells, and repair damaged brain cells. However, the clinical effects of add-on Astragalus in improving cognition in these patients remain unclear. Therefore, this pragmatic clinical trial aims to determine the efficacy and safety of add-on Astragalus in improving cognition in patients with AD

ELIGIBILITY:
Inclusion Criteria:

1. Participate voluntarily and sign an informed consent form
2. Age 50-85 years old;
3. Memory loss for at least 6 months with a tendency of progressive deterioration;
4. Mild or moderate patients, i.e. MMSE total score:14< MMSE total score<24, 0.5≤CDR-GS≤2;
5. The highest likelihood of AD (medial temporal lobe atrophy visual rating scale grade 2 or higher on coronal imaging) as demonstrated by cranial MRI scanning and oblique coronal hippocampal scanning review at the time of screening;
6. Hachinski Ischemia Scale (HIS) score < 4;
7. A diagnosis of dementia according to the DSM-V and a diagnosis of "probable AD" according to the NIA-AA criteria;
8. No significant positive signs on neurological examination;
9. The subject has the ability to read, write, and communicate, the subject has a stable and reliable caregiver or at least has frequent contact with the caregiver (at least 2 hours per day, 4 days per week), the caregiver will help the patient to participate in the study, the caregiver must accompany the subject to the study visit, and there must be sufficient interaction with the subject to provide valuable information for the rating of the scales. information for each scale score;
10. The underlying treatment for AD prior to enrolment remains unchanged, but needs to have been on long-term stable use for more than 4 weeks prior to randomisation to the subgroups, and the dose remains stable during the study period. Such drugs include:cholinesterase inhibitors and memantine;
11. The TCM diagnosis was spleen and kidney deficiency. -

Exclusion Criteria:

1. Non-AD-induced memory and cognitive impairment, such as a diagnosis of other types of dementia, including, but not limited to, Mixed Disease Dementia, Vascular Dementia, Parkinson's Disease Dementia, Lewy Body Dementia, Huntington's Chorea-related Dementia, Normal Pressure Hydrocephalus, Brain Tumour, Progressive Supranuclear Palsy, Frontotemporal Lobar Dementia, etc.; Endocrine system pathology (e.g., Thyroid Disease, Parathyroid Disease) as well as Folic Acid, Vitamin B12 deficiency or any other causes of dementia; the presence of impaired consciousness, etc;
2. A history of seizures; psychosis, including but not limited to schizophrenia, schizoaffective disorder, bipolar disorder, or delirium; and
3. Hamilton Depression Scale (HAMD) score >17;
4. Significant focal lesions on MRI with one of the following: a. >2 infarct foci >2cm in diameter; b. Infarct foci in key areas such as thalamus, hippocampus, internal olfactory cortex, parafrontal olfactory cortex, angular gyrus, cortex, and other subcortical grey matter nuclei; and c. Cerebral white matter damage with a Fazekas Scale score ≥3;
5. Patients who have taken other herbal preparations within the past 1 month;
6. Astragalus allergy or contraindication;
7. Presence of abnormal laboratory parameters: impaired renal function (blood Cr > 1.5xULN) or creatinine clearance (C cr) < 50mL/min or abnormal liver function (ALT or AST > 2xULN);
8. Patients who refused or had contraindications to MRI or EEG (pacemakers, coronary and peripheral arterial stents, metallic implants, claustrophobia, or severe visual or hearing impairments); refused to have blood drawn;
9. Hachinski Ischaemia Scale score ≥ 4;
10. Pregnant or breastfeeding patients; and
11. Other unmanageable clinical problems (e.g. neoplasms, HIV infection, syphilis spirochete infection, hepatitis C virus infection, active hepatitis B or other severe chronic infectious diseases, severe neurological, cardiovascular, respiratory and other systemic diseases);
12. Patients who have participated in other clinical studies within the past 3 months;
13. Those who, in the opinion of the investigator, need to be excluded

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcome measure will be the absolute change in the Clinical Dementia Rating | Participants were followed up for 24 weeks after baseline.
  Clinical Dementia Rating scale scores range from 0 to 18, with higher scores indicating worse.

SECONDARY OUTCOMES:
The absolute scores change in the Rey-Osterrieth Complex Figure Test [ROCF] recall score between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  The ROCF scale scores range from 0 to 36, with higher scores indicating better.
The absolute scores change in the Rey-Osterrieth Complex Figure Test-copy score between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  The ROCF copy scale scores range from 0 to 36, with higher scores indicating better.
The absolute scores change in the Trail Making Test-A score between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  The Trail Making Test-A scores range from 0 to 25, with higher scores indicating better.
The absolute scores change in the Digit Span Forward score between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  TheDigit Span Forward score scores range from 0 to 10, with higher scores indicating better.
The absolute scores change in the Trail Making Test-B score between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  The Trail Making Test-B scores range from 0 to 25, with higher scores indicating better.
The absolute scores change in the Digit Span Backward score between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  The Digit Span Forward score scores range from 0 to 9, with higher scores indicating better.
The absolute scores change in the Verbal Fluency Test score between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  The Verbal Fluency Test score scores range from 0 to 14, with higher scores indicating better.
The absolute scores change in the Hamilton Anxiety Scale score between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  The Hamilton Anxiety Scale score scores range from 0 to 56, with higher scores indicating worse.
The absolute scores change in the Hamilton Depression Scale score between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  The Hamilton Anxiety Scale score scores range from 0 to 96, with higher scores indicating worse
The absolute change in the blood pressure between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  To observe the changes of orthostatic blood pressure in patients
The absolute change in the level of plasma β-amyloid40 (ng/ml) between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  Amyloid is one of the main biomarkers of dementia
The absolute change in the level of plasma β-amyloid42 (ng/ml) between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  Amyloid is one of the main biomarkers of dementia
The absolute change in the level of plasma glial fibrillary acidic protein (ng/ml) between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  Glial fibrillary acidic protein is one of the main biomarkers of dementia
The absolute change in the level of plasma neurofilament light chain (ng/ml) between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  Neurofilament light chain is one of the main biomarkers of dementia
The absolute change in the level of plasma hyper-phosphorylated tau-181 (ng/ml) between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  Neurofilament light chain is one of the main biomarkers of dementia
The absolute change in the neurite density index between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  Neurite density index, range from 0-1, is the main indicator of neurite-oriented diffusion and density imaging (NODDI),with higher scores indicating better
The absolute change in the orientation dispersion index between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  Orientation dispersion indexrange from 0-1, is the main indicator of neurite-oriented diffusion and density imaging (NODDI) ,with higher scores indicating better.
The absolute change in the isotropic volume fraction between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  Isotropic volume fraction, range from 0-1, is the main indicator of neurite-oriented diffusion and density imaging (NODDI), with higher scores indicating worse .
The absolute change in thickness, between baseline and week 24. | Participants were followed up for 24 weeks after baseline.
  Cortical thickness is the main indicator of grey matter.Cortical thickness was obtained by analyzing structural MRI using the freesurfer.
The absolute change in volume, between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  Volume, is the main indicator of brain structure.Volume was obtained by analyzing structural MRI using thevoxel-based morphometry
The absolute change in delta, between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  Delta, is the main indicator of the cerebral cortex activity
The absolute change in theta, between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  Theta, is the main indicator of the cerebral cortex activity（range from 4-7.5Hz）
The absolute change in alpha, between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  Alpha, is the main indicator of the cerebral cortex activity（range from 7.5-14Hz）
The absolute change in beta1, between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  Beta1, is the main indicator of the cerebral cortex activity（range from 14-20Hz）
The absolute change in beta2, between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  Beta2, is the main indicator of the cerebral cortex activity（range from 20-30Hz）
The absolute change in gamma, between baseline and week 24 | Participants were followed up for 24 weeks after baseline.
  Gamma, is the main indicator of the cerebral cortex activity（range from 30-50Hz）

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No